CLINICAL TRIAL: NCT00128986
Title: A Phase I Study of Tomotherapy in Patients With Benign Brain Tumour
Brief Title: Study of Tomotherapy in Patients With Benign Brain Tumour
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNS-09-0029 / ethics 21879
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Brain Neoplasms
Keywords: radiotherapy; brain
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Tomotherapy — 3T MRS scans (3T magnetic resonance spectroscopy)

SUMMARY:
Although malignant brain tumors are the most common type of primary brain tumor, there are a number of other benign brain tumors that exist. Many difficulties exist with treating these tumors that have led to controversies in the best treatment. A common issue among these brain tumors is the risk of long term side effects from treatment. What limits the use of curative radiation therapy is the ability to deliver a maximal dose to the tumor while minimizing the amount of radiation to the normal structures in the brain. A new method of delivering radiation, called tomotherapy, has been acquired at the Cross Cancer Institute (CCI) and will be used in this study. It has the ability to deliver a high dose of radiation to the tumor while minimizing the amount of radiation to normal brain structures. This study will use this method of radiation therapy to deliver radiation and see if the long term side effects from radiation therapy can be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed newly diagnosed base of skull benign tumour
* Karnofsky Performance Status (KPS) equal to or greater than 70

Exclusion Criteria:

* Brain metastases or recurrent tumour
* Prior radiotherapy (RT) to head or neck
* No prior chemotherapy or radiosensitizer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
safety and adverse effects | Trial Completion

SECONDARY OUTCOMES:
efficacy and survival | Trial completion

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Roa, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada